# Extension Study in a Cohort of Adult Patients With SARS-CoV-2 Infection Requiring Hospital Admission and Received Treatment With Plitidepsin in the APLICOV-PC Study

Statistical Analysis Plan

NCT05121740

November 17, 2022



# E-APLICOV-PC (AV-APL-A-003-21)

Extension study in a cohort of adult patients with SARS-CoV-2 infection requiring hospital admission who received treatment with plitidepsin in the APLICOV-PC.

## STATISTICAL ANALYSIS PLAN

Version: 2.0

Date: 17-NOV-2022

# **Table of contents**

| 1 | Int | roduction | 3 |
|----|------|------------------------------------------------------|----|
| 2 | Sy | nopsis | 4 |
| | 2.1 | Title of the study | 4 |
| | 2.2 | Justification of the study | 4 |
| | 2.3 | Code of the study | 5 |
| | 2.4 | Sponsor | 5 |
| | 2.5 | Design | 5 |
| | 2.6 | Study Objectives | 5 |
| | 2.7 | Endpoints | 5 |
| | 2.8 | Study population | 5 |
| | 2.9 | Inclusion criteria | 6 |
| | 2.10 | Exclusion criteria | 6 |
| 3 | Ge | eneral principles | 6 |
| 4 | lm | putation | 6 |
| 5 | St | udy analysis populations | 6 |
| | 5.1 | Definition of the study population to be analyzed | 7 |
| | 5.2 | Patients disposition | 7 |
| | 5.3 | End of treatment | 7 |
| | 5.4 | End of study | 7 |
| | 5.5 | Deaths | 7 |
| 6 | Pa | atients description | 7 |
| | 6.1 | Demographic data description. General considerations | 7 |
| | 6.2 | Patients characteristics | 7 |
| 7 | An | nalysis of the primary endpoint | 8 |
| 8 | Ot | her analysis | 9 |
| 9 | Lis | sting | 10 |
| 1( | ) | Study population | 12 |
| 1 | 1 | Primary endpoints | 14 |
| 12 | 2 | Other analysis | 23 |
| 1: | 3 | Other Listings | 31 |
| 14 | 4 | ICH Listings | 32 |
| 1 | 5 | History of changes | 33 |

## 1 Introduction

This statistical analysis plan describes the protocol-defined final analysis that will be performed in the E-APLICOV-PC study (AV-APL-A-003-21).

## **Abbreviations:**

| Abbreviation | Term |
|--------------|----------------------------------------------|
| AE | Adverse event |
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| ATC | Anatomical therapeutic chemical |
| BMI | Body mass index |
| bpm | Beats per minute |
| BSA | Body surface area |
| °C | Degrees Celsius |
| cm | Centimeter/s |
| COVID-19 | Coronavirus disease 2019 |
| CPK | Creatine phosphokinase |
| DBP | Diastolic blood pressure |
| ECG | Electrocardiogram |
| ЕСНО | Echocardiogram |
| eCRF | Electronic case report form |
| $FEV_1$ | Forced expiratory volume in 1 second |
| FVC | Forced vital capacity |
| ICH | International conference on harmonization |
| G1-X | Grade 1-X |
| GGT | Gamma-glutamyl transferase |
| HR | Heart rate |
| ICU | Intensive care unit |
| id. | Identifier |
| i.e. | That is, from Latin id est |
| IgG | Immunoglobulin G |
| Kg | Kilogram/s |
| LDH | Lactate dehydrogenase |
| MedDRA | Medical dictionary for regulatory activities |
| m | Meter/s |
| mg | Milligram/s |
| mmHg | Millimeter of mercury |

mMRC Modified medical research council

ms milliseconds

MUGA Multigated acquisition scan

6MWT Six-minute walk test

N Number

NCI-CTCAE National Cancer Institute-Common Terminology Criteria for

Adverse Events

PaFi

(PAO<sub>2</sub>/FiO<sub>2</sub>) Ratio of partial pressure arterial oxygen and fraction of inspired

Ratio oxygen

PCR Polymerase chain reaction

PR PR interval
PT Preferred term
Q1 First quartile
Q3 Third quartile
QT QT interval

RR Respiratory rate

SAE Serious adverse event SaO<sub>2</sub> Oxygen saturation

SARS-CoV-2 Severe acute respiratory syndrome coronavirus 2

SAS Statistical analysis system
SAEs Serious adverse events
SBP Systolic blood pressure
SOC System organ classes
Std Standard deviation
ULN Upper limit of normal

WHO World health organization

WBC White blood cell

## 2 Synopsis

## 2.1 Title of the study

Extension study in a cohort of adult patients with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection requiring hospital admission who received treatment with plitidepsin in the APLICOV-PC.

### 2.2 Justification of the study

The APLICOV-PC proof of concept study demonstrated the antiviral activity of plitidepsin in terms of viral load reduction, recovery induction, lymphocyte and other inflammatory parameters reconstitution.

Approximately 10 to 25% of patients with COVID-19 experience symptoms beyond 3 months, resulting in a significant restriction in their everyday lives due to the sequelae of the disease that may persist for a year or more and entail long-term medical leaves.

The aim of this study is to assess whether the treatment with plitidepsin, by attaining a reduction in the viral load and a faster recovery of the patient, could have a relevant impact in preventing the appearance of sequelae resulting from the SARS-CoV-2 infection.

### 2.3 Code of the study

E-APLICOV-PC (AV-APL-A-003-21).

## 2.4 Sponsor

Pharma Mar, S.A

## 25 Design

Multi-site extension study of the APLICOV-PC clinical study follow-up.

To participate in the study, the patients must have previously participated in the APLICOV-PC proof of concept study and may have received:

- 1.5 mg of plitidepsin administered as a 1.5-hour infusion, once a day for 3 consecutive days (total dose 4.5 mg).
- 2.0 mg of plitidepsin administered as a 1.5-hour infusion, once a day for 3 consecutive days (total dose 6.0 mg).
- 2.5 mg of plitidepsin administered as a 1.5-hour infusion, once a day for 3 consecutive days (total dose 7.5 mg).

Patients were enrolled after signing informed consent to participate in this extension study.

## 2.6 Study Objectives

To evaluate the incidence of post-COVID-19 morbidity and characterize the profile of complications in patients who participated in the APLICOV-PC study.

#### 2.7 Endpoints

Incidence of post-COVID-19 complications.

### 2.8 Study population

The main objective of the study is to evaluate the incidence of post-COVID-19 morbidity and

characterize the profile of complications in patients who participated in the APLICOV-PC study. The maximum number of patients who can participate in the trial is limited to 42.

#### 2.9 Inclusion criteria

Patient who participated in the APLICOV-PC study treated with plitidepsin and who gives their consent.

#### 2.10 Exclusion criteria

There are no exclusion criteria for this study.

## 3 General principles

Planned analyses in this document will be carried out once the database is declared cleaned, closed and approved by Pharma Mar according to the premises described in the Data Management Plan version 1.0 approved on 12-Jan-2022.

Statistical analyses will be performed using Statistical Analysis System (SAS) software version 9.4 and RStudio. The results of the analyses will be presented in editable format (i.e. rtf).

The data will be provided with one decimal place in general. In those cases where greater precision is required, as many decimal places as necessary will be provided.

Before performing the analysis, the following terms should be coded/reviewed and approved:

- Adverse events (AEs), hospital readmissions and COVID-19 complications. Coded according to Medical Dictionary for Regulatory Activities (MedDRA) and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.
- Medication. Classified according to the WhoDrug dictionary (latest version available).
- Reconciliation between the clinical database and the Pharmacovigilance database of serious adverse events (SAEs) in the study, including the resolution of all discrepancies.

Analysis will be done separately for each arm and the total population.

Continuous variables will be presented through the mean, median, standard deviation, range, first quartile (Q1) and third quartile (Q3). Categorical variables will be displayed through the distribution of frequencies and percentages; percentages with valid data will be presented and missing values will not be taken into account in the percentage calculation.

## 4 Imputation

There is no strategies/methods to handle missing data.

## 5 Study analysis populations

#### 5.1 Definition of the study population to be analyzed

All patients who sign an informed consent form and agree to undergo the set of clinical examinations, imaging and laboratory tests specified in section 10 of the protocol, will be analyzed in order to fulfil the objectives of the study.

### 5.2 Patients disposition

The number and percentage of patients per center will be provided.

All analysis will be performed separately for each arm and a total column will be added.

#### 53 End of treatment

There is no end of treatment for this study as no treatment doses are administered.

### 5.4 End of study

The number and percentage of patients who completed or not the study will be provided. For those patients who finished the study early, the causes of termination will be described. The cases considered as early termination are:

- Withdrawal of consent
- Follow up completed
- Lost to follow-up
- Death
- Other

All analysis will be performed separately for each arm and a total column will be added.

#### 55 Deaths

The number and percentage of patients who died during the study will be provided. Patients who have died due to an AE will be described in more detail, indicating all the variables related to the AEs registered in the electronic case report form (eCRF).

All the analyses will be performed separately for each arm and a total column will be added.

## 6 Patients description

#### 6.1 Demographic data description. General considerations.

The characteristics of the patients will be described and the unavailable information will be detailed; not available values will not be taken into account in the percentage calculation, only valid percentages will be presented. The analysis will be carried out on the full population and all results will be provided by treatment arm. Aggregated results as well as patient listings will be provided.

#### 6.2 Patients characteristics

Demographic and baseline data:

- Age (years)
- Gender (male/female)
- Ethnic group (Arab; Caucasian; Latin; Asian; Black; Other)
- Weight (kg)
- Height (cm)
- Body surface area (BSA) (m<sup>2</sup>)
- Body mass index (BMI) calculated

In addition to all the basal characteristics used in APLICOV-PC if it necessary.

## 7 Analysis of the primary endpoint

The main objective of the study is to evaluate the incidence of post-COVID-19 morbidity and characterize the profile of complications in the cohort of patients who participated in the APLICOV-PC study.

The number and percentage of patients who develop complications related to persistent illness, according to the physician, during the period between the end of the APLICOV-PC proof of concept study and the completion of this extension study by the patient, as well as the percentage of patients who present complications will be detailed.

A description of the following endpoints will be presented:

- Number and percentage of patients who required readmission to hospital and causes, since last visit of APLICOV-PC study until the end of this extension study.
- Number and percentage of patients who needed oxygen therapy and duration of the same, since last visit of APLICOV-PC study until the end of this extension study.
- The maximum, minimum, Q1 and Q3, mean, median and standard deviation (Std) of the duration of the oxygen therapy.
- Number and percentage of patients who presented complications (defined in Annex 5 of the protocol).
- Barthel Index. A description with the frequency and percentage of each dependency category, according to the score obtained, will be provided:
  - 0-20: Total dependency
  - 21-60: Severe dependency
  - 61-90: Moderate dependency
  - 91-99: Slight dependency
  - 100: Independence
- The maximum, minimum, Q1 and Q3, mean, median and Std of the parameters related to pulmonary function will be provided: oxygen saturation (SaO<sub>2</sub>), ratio of partial pressure arterial oxygen and fraction of inspired oxygen (PAFI), forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1), FEV1/FVC and diffusion test.

- The maximum, minimum, Q1 and Q3, mean, median and Std of the results of the Sixminute walk test (6MWT).
- Frequency and percentage of each category of the modified Medical Research Council (mMRC) scale:
  - 0 (Dyspnea only after strenuous exercise)
  - 1 (Dyspnea occurring when hurrying on level ground or walking up a slight incline)
  - 2 (Dyspnea resulting in walking more slowly than people of the same age on level ground or in stopping for breath when walking at own pace on level ground)
  - 3 (Dyspnea resulting in stopping for breath after walking about 100 meters of after a few minutes on level ground)
  - 4 (Dyspnea severe enough to prevent the person from leaving the house or occurring when dressing or undressing)
- In patients who present pneumonia upon entry into the APLICOV-PC study, number and percentage of patients with abnormalities in the chest X-ray and description of these abnormalities.
- Number and percentage of patients who presented abnormalities  $\geq$ G2 in the analytical parameters.
- Number and percentage of patients who presented abnormalities in the electrocardiogram (ECG) and description of these abnormalities.
- In patients suffering a relevant cardiac event during their participation in the APLICOV-PC study, number and percentage of patients who presented abnormalities in the heart Ultrasound/multigated acquisition scan (MUGA) and description of these abnormalities.
- Multivariate analysis to evaluate the relationship of the main covariates in the previous study (APLICOV-PC). More relevant exploratory covariates from the univariate analyses (p-value < 0.10) will be included in the multivariate analyses. The endpoints listed were correlated with the patients' basal characteristics, the degree of severity of the illness, comorbidities, the plitidepsin dosage, the viral load and the clinical evolution documented in the APLICOV-PC study.

## 8 Other analysis

- The maximum, minimum, Q1 and Q3, mean, median and Std of the vital signs will be provided: systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR), temperature and respiratory rate.
- The maximum, minimum, Q1 and Q3, mean, median and Std of ECG parameters.
- Number and percentage of patients with abnormalities in the physical examination. The result will be listed.
- Number and percentage of patients with abnormalities in the neurological examination. The result will be listed.
- A description will be provided with the frequency and percentage of each category of the lung diffusion test:
  - Normal (between the 80 % and 120 % of the reference value)
  - Low (below the 80 % of the reference value)

- High (over the 120 % of the reference value)
- Number and percentage of patients who have been diagnosed of COVID-19 since the completion of APLICOV-PC study.
- Number and percentage of patients who have received any COVID-19 vaccine and the number of doses.
- Number and percentage of related or unknown post-COVID-19 complication. Worst per patient.
- Number and percentage of all post-COVID-19 complications. Worst grade per patient.
- Number and percentage of related post-COVID-19 complications. Worst grade per patient.
- Number and percentage of patients with at least AE.
- Number and percentage of patients with at least SAE.
- Number and percentage of patients with at least grade  $\geq$  3 AE.
- Number and percentage of patients with AEs by system organ classes (SOC) and preferred term (PT), regardless of relationship.
- The maximum, minimum, Q1 and Q3, mean, median and Std of laboratory parameters.
- Aplicov-pc summay of Demographic and Other Baseline Characteristics table of patients include in this study by dose and severity of disease.
  - o Median (range) time from symptom onset to first plitidepsin administration, days
  - o Number of comorbidities, n (%) (none, one, two or more)
  - Comorbidities, n (%) (Cardiac disease, Kidney disease, Liver disease, Lung disease (COPD), Asthma, Diabetes, Hypertension, Obesity)
  - Clinical status at randomization, n (%)
  - Vital signs, median (range) (Body temperature, °C, Systolic blood pressure, mmHg,
  - o Diastolic blood pressure, mmHg, Heart rate, bpm, Respiratory rate, bpm, SpO2
  - o B, %, On oxygen at baseline, n (%))
  - Laboratory parameters, median (range) (WBC, x109/L, Platelet count, x109/L, Lymphocytes, x109/L, Serum creatinine, μmol/L, ALT x ULN, AST x ULN, LDH x ULN, CPK x ULN, GGT x ULN, C-reactive protein, Ferritin, D-dimer)
  - o log10 copies/mL viral load, median (range)
  - o Days from Plitidepsin to first complication
  - Days from hospital discharge to first complication
  - o Time from Plitidipesin first-dose to E-APLICOV inclusion (Month)

## 9 Listing

- Post-COVID-19 complications will be listed.
- Hospital readmission will be listed
- Oxygen therapy will be listed
- The medication administered before starting the 6MWT will be listed.
- The results of the ECG will be listed.

- The results of the chest X-ray will be listed.
- The ECHO/MUGA results will be listed
- The hematological laboratory parameters will be listed.
- The coagulation laboratory parameters will be listed.
- The biochemistry laboratory parameters will be listed.
- The pharmacological treatments will be listed
- The AEs will be listed
- Physical examination will be listed
- The neurological examination will be listed
- The vaccination schedule will be listed
- The COVID-19 (PCR) will be listed
- The COVID-19 history will be listed
- The serology SARS-CoV-2 will be listed

# Appendix I

# 10 Study population

Table 10.1 Analyzed patients

| | Dose Cohort | | |
|---|---|---|---|
| | 1.5 mg 2.0 mg 2.5 mg Tot N=X N=X N= | | |
| | | n (% | 5) |
| Analyzed patients | | | |

Table 10.2 Subject Disposition by site

| | | Dose Cohort | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Sites | 1.5 | mg | 2.0 | ) mg | 2.5 | mg | Total | |
| | N= | =X | N: | =X | N= | =X | N=X | |
| | | | | n ( | n (%) | | | |
| | Recruited | Recruited Analyzed | | Analyzed | Recruited | Analyzed | Recruited | Analyzed |
| Site 1 | | | | | | | | |
| Site 2 | | | | | | | | |
| Site | | | | | | | | |

Table 10.3 End of study

| | Dose Cohort | | | |
|---|---|---|---|---|
| | 1.5 mg<br>N=X | 2.0 mg<br>N=X | 2.5 mg<br>N=X | Total<br>N=X |
| | | n (% | 5) | |
| End of study reasons | | | | |
| Follow-up completed as per protocol | | | | |
| Lost to follow-up | | | | |
| Withdrawal of consent | | | | |
| Death | | | | |
| Other | | | | |

Table 10.4 Demographics (categorical)

| | | Dose Cohort | |
|---|---|---|---|
| | 1.5 mg<br>N=X | 1.5 mg 2.0 mg 2.5 mg N=X N=X | |
| | | n (% | (a) |
| Gender | | | |
| Ethnic group | | | |

Table 10.5 Demographics (Continuous)

| | | Dose Cohort | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Continuous endpoints | 1.5 | | | | | | Total | | | | | | |
| | N | Mean | Median | Range | Q1 | * | | N | Mean | Median | Range | Q1 | * |
| Age | | | | | | | | | | | | | |
| Weight (kg) | | | | | | | | | | | | | |
| Height (cm) | | | | | | | | | | | | | |
| BSA (m²) | | | | | | | | | | | | | |
| BMI | | | | | | | | | | | | | |

<sup>\*</sup> Q3 and Std.

# Appendix II

# 11 Primary endpoints

Table 11.1.1 End points I by dose cohort

| | | Dose | Cohort | |
|---|---|---|---|---|
| Endpoints | 1.5 mg<br>N=X | 2.0 mg<br>N=X | 2.5 mg<br>N=X | Total<br>N=X |
| | | n ( | (%) | |
| Patients who presented post-<br>COVID-19 complications<br>(related or unknown<br>relationship to study disease) | | | | |
| Patients who presented post-<br>COVID-19 complications<br>(regardless relationship) | | | | |
| Patients who presented post-<br>COVID-19 complications<br>(related to study disease) | | | | |
| Patients who required readmission to hospital (regardless of relationship) | | | | |
| Patients who required readmission to hospital (COVID-19) | | | | |
| Patients who required readmission to hospital (post COVID-19 complication) | | | | |
| Patients who required oxygen therapy | | | | |
| Patients with abnormalities in the chest X-ray* | | | | |
| Patients who presented abnormalities ≥G2 in the analytical parameters | | | | |
| Patients who presented abnormalities in the ECG | | | | |
| Patients who presented abnormalities in the heart Ultrasound/MUGA** | | minte the ADLIC | | |

Table 11.1.2 End points I by Severity of disease

| | | Severity of | of disease | |
|-----------|-------------|-----------------|---------------|--------------|
| Endpoints | Mild<br>N=X | Moderate<br>N=X | Severe<br>N=X | Total<br>N=X |

<sup>\*</sup>Only in patients who present pneumonia upon entry into the APLICOV-PC

\*\* Only in patients who suffered a relevant cardiac event during their participation in the APLICOV-PC study

| D. C. 1 1 1 1 | |
|--------------------------------|------|
| Patients who presented post- | |
| COVID-19 complications | |
| (related or unknown | |
| relationship to study disease) | |
| Patients who presented post- | |
| COVID-19 complications | |
| (regardless relationship) | |
| Patients who presented post- | |
| COVID-19 complications | |
| (related to study disease) | |
| Patients who required | |
| readmission to hospital | |
| (regardless of relationship) | |
| Patients who required | |
| readmission to hospital | |
| (COVID-19) | |
| Patients who required | |
| readmission to hospital | |
| (post COVID-19 | |
| complication) | |
| Patients who required oxygen | |
| therapy | |
| Patients with abnormalities in | <br> |
| the chest X-ray* | _ |
| Patients who presented | |
| abnormalities ≥G2 in the | |
| analytical parameters | |
| Patients who presented | |
| abnormalities in the ECG | |
| Patients who presented | |
| abnormalities in the heart | |
| Ultrasound/MUGA** | |

Table 11.2.1.1 Summary of post-COVID-19 complications, regardless of relationship, by dose cohort and overall. Worst per patient

| | | Dose Cohort | | |
|---|---|---|---|---|
| Post COVID 10 complications | 1.5 mg | 2.0 mg | 2.5 mg | Total |
| Post-COVID-19 complications | N=X | N=X | N=X | N=X |
| | | n ( | (%) | |
| Asthenia | | | | |
| General discomfort | | | | |

Table 11.2.1.2 Summary of post-COVID-19 complications, regardless of relationship, by severity of disease and overall. Worst per patient

| | Severity of disease | | | |
|---|---|---|---|---|
| Post-COVID-19 complications | Mild | Moderate | Severe | Total |
| r r | N=X | N=X | N=X | N=X |
| | | n (° | %) | |

<sup>\*</sup>Only in patients who present pneumonia upon entry into the APLICOV-PC

\*\* Only in patients who suffered a relevant cardiac event during their participation in the APLICOV-PC study

| Anxiety |
|----------|
| Asthenia |

Table 11.2.2 Summary of Complications, Related to study disease, by dose cohort and overall

| | | Dose | Cohort | |
|-----------------------------|--------|--------|--------|-------|
| Post-COVID-19 complications | 1.5 mg | 2.0 mg | 2.5 mg | Total |
| Fost-COVID-19 complications | N=X | N=X | N=X | N=X |
| | | n ( | (%) | |
| Asthenia | | | | |
| General discomfort | | | | |

Table 11.3.1 Summary of post-COVID-19 complications, by grade and overall. Worst grade per patient. (Dose  $1.5\ / 2\ / 2.5\ mg$  and total)

| | | ( | G1 | | G2 | ( | <del>3</del> 3 | | •• | Te | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | N | % | N | % | N | % | N | % | N | % |
| Post-COVID-19 | Asthenia | | | | | | | | | | |
| complications | | | | | | | | | | | |

Table 11.3.2 Summary of post-COVID-19 complications, related to study disease, by grade and overall. Worst grade per patient. (Dose 1.5 / 2 / 2.5 mg and total)

| | | ( | G1 | | G2 | ( | 33 | | | To | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | N | % | N | % | N | % | N | % | N | % |
| Post-COVID-19 complications | Asthenia | | | | | | | | | | |
| complications | | | | | | | | | | | |

Listing 11.1.1 Post-COVID-19 complications

| Dose<br>cohort | Subject id. | Post-<br>COVID-19<br>complication | Start<br>date | End<br>date | Ongoing | Duration. | First Date<br>Plitidepsin<br>dose | Relationship | Severity<br>of disease |
|---|---|---|---|---|---|---|---|---|---|

Listing 11.1.2 Post-COVID-19 complications (related to study disease)

| Dose cohort | Subject id. | Post-<br>COVID-19<br>complication | Start<br>date | End<br>date | Ongoing | First Date<br>Plitidepsin<br>dose | Relationship | Severity<br>of disease |
|---|---|---|---|---|---|---|---|---|

Table 11.4 Post-COVID-19 complications duration

| | | | | | | | Do | ose ( | Coh | ort | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Continuous endpoints | | | 1.5 | | | | | ••• | | | | | Tota | al | | |
| | N | Mean | Median | Range | Q1 | * | <br> | | | | <br>N | Mean | Median | Range | Q1 | * |
| Post-COVID-<br>19<br>complications<br>duration | | | | | | | | | | | | | | | | |
| Asthenia | | | | | | | | | | | | | | | | |

<sup>\*</sup> Q3 and Std.

Listing 11.2 Hospital readmission

| Dose cohort | Subject id. | Hospital readmission | Reason | ICU admission | Start<br>date | End<br>date | Ongoing | Duration |
|---|---|---|---|---|---|---|---|---|

Table 11.5 Oxygen therapy duration

| | | | | | | | D | ose | Coh | ort | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Continuous endpoints | | | | 1.5 | | | | | | | | | | Tot | al | | |
| | N | Mean | Median | Range | Q1 | * | | | | | <br> | N | Mean | Median | Range | Q1 | * |
| Oxygen<br>therapy<br>duration | | | | | | | | | | | | | | | | | |
| Type** | | | | | | | | | | | | | | | | | |

<sup>\*</sup> Q3 and Std.

\*\*Nasal cannula; Simple face mask; Venturi mask; Non-rebreather mask; Invasive mechanical ventilation (IMV); Other, specify

Listing 11.3 Oxygen therapy required

| Dose | Subject id. | Oxygen<br>therapy<br>required | Туре | Start date | End date | Ongoing | Duration |
|---|---|---|---|---|---|---|---|

Table 11.6 Pulmonary function assessment and diffusion test

| | | | | | | | Do | ose | Col | nort | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Continuous endpoints | | | 1.: | 5 | | | | | | | | | Tota | ıl | | |
| | N | Mean | Median | Range | Q1 | * | <br> | | | | <br>N | Mean | Median | Range | Q1 | * |
| Pulmonary<br>function<br>assessment | | | | | | | | | | | | | | | | |
| SaO <sub>2</sub> (%) | | | | | | | | | | | | | | | | |
| PAO <sub>2</sub> /FiO <sub>2</sub> | | | | | | | | | | | | | | | | |
| Spirometry | | | | | | | | | | | | | | | | |
| FVC (ml) | | | | | | | | | | | | | | | | |
| FEV1(ml) | | | | | | | | | | | | | | | | |
| FEV1 /FVC | | | | | | | | | | | | | | | | |
| Lung diffusion reference theoretical value | | | | | | | | | | | | | | | | |

<sup>\*</sup> Q3 and Std.

Table 11.7 Pulmonary function assessment

| | | Dose | Cohort | |
|------------------------|--------|--------|--------|-------|
| | 1.5 mg | 2.0 mg | 2.5 mg | Total |
| | N=X | N=X | N=X | N=X |
| | | n ( | (%) | |
| Spirometry | | | | |
| Normal (≥80%) | | | | |
| Reduced (<80%) | | | | |
| Lung diffusion testing | | | | |
| Normal | | | | |
| Low | | | | |
| High | | | | |

| Dyspnea assessment (mMRC) |
|---------------------------|
| 0 |
| 1 |
| 2 |
| 3 |
| 4 |

Table 11.8 Barthel scale

| | | Dose | Cohort | |
|---------------------------|--------|--------|--------|-------|
| | 1.5 mg | 2.0 mg | 2.5 mg | Total |
| | N=X | N=X | N=X | N=X |
| | | n ( | %) | |
| Barthel scale | | | | |
| Total dependency (0-20) | | | | |
| Severe dependency (21-60) | | | | |
| Moderate | | | | |
| dependency (61-90) | | | | |
| Slight dependency (91-99) | | | | |
| Independence (100) | | | | |

Table 11.9 Six-minute walk test (I)

| | Dose Cohort | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Continuous endpoints- 6MWT | 1.5 | | | | | | Tot | tal | | | | | |
| | N | Mean | Median | Range | Q1 | * | | N | Mean | Median | Range | Q1 | * |
| Pre-TEST | | | | | | | | | | | | | |
| Weigth (Kg) | | | | | | | | | | | | | |
| SBP (mmHg) | | | | | | | | | | | | | |
| DBP (mmHg) | | | | | | | | | | | | | |
| SpO <sub>2</sub> (%) | | | | | | | | | | | | | |
| Heart rate (bpm) | | | | | | | | | | | | | |
| Post-TEST | | | | | | | | | | | | | |
| SpO <sub>2</sub> (%) | | | | | | | | | | | | | |
| Heart rate (bpm) | | | | | | | | | | | | | |
| Results | | | | | | | | | | | | | |

| | Dose Cohort | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Continuous endpoints- 6MWT | | 1.5 | | | | | Total | | | | | | | |
| | N | Mean | Median | Range | Q1 | * | | <br> | N | Mean | Median | Range | Q1 | * |
| Total distance (m) | | | | | | | | | | | | | | |
| Expected distance | | | | | | | | | | | | | | |
| (m) | | | | | | | | | | | | | | |
| Expected percentage | | | | | | | | | | | | | | |
| (m) | | | | | | | | | | | | | | |
| Nº laps | | | | | | | | | | | | | | |

<sup>\*</sup> Q3 and Std.

Table 11.10.1 Six-minute walk test (II) by dose cohort

| | | Dose ( | Cohort | |
|---|---|---|---|---|
| Categorical Endpoints (6MWT) | 1.5 mg<br>N=X | 2.0 mg<br>N=X | 2.5 mg<br>N=X | Total<br>N=X |
| | | n ( | %) | |
| Pre-TEST | | | | |
| Borg scale of dyspnea and fatigue at basal (1): | | | | |
| Post-TEST | | | | |
| Borg scale of dyspnea and fatigue after test (1): | | | | |
| Results | | | | |
| Stopped or paused | | | | |
| Other symptoms at the end of the exercise (2) | | | | |

<sup>(1) 0 (</sup>None); 0.5 (Very, very slight), 1 (Very slight); 2 (Slight); 3 (Moderate); 4 (Somewhat severe); 5 (Severe); 6 (Severe); 7 (Very severe); 8 (Very severe); 9 (Very very severe); 10 (Maximal).

Table 11.10.2 Six-minute walk test (II) by severity of disease

| | | Severity of | of disease | |
|---|---|---|---|---|
| Categorical Endpoints (6MWT) | Mild | Moderate | Severe | Total |
| | N=X | N=X | N=X | N=X |
| | | n (' | %) | |
| Pre-TEST | | | | |
| Borg scale of dyspnea and fatigue at basal (1): | | | | |
| Post-TEST | | | | |
| Borg scale of dyspnea and fatigue after test (1): | | | | |
| Results | | | | |
| Stopped or paused | | | | |

<sup>(2)</sup> Angina; Dizziness; Pain in hip, leg or calf; None

| Other symptoms at the end of the exercise (2) |
|-----------------------------------------------|

<sup>(1) 0 (</sup>None); 0.5 (Very, very slight), 1 (Very slight); 2 (Slight); 3 (Moderate); 4 (Somewhat severe); 5 (Severe); 6 (Severe); 7 (Very severe); 8 (Very severe); 9 (Very very severe); 10 (Maximal).

## Listing 11.4 Abnormalities in the chest X-ray

| Dose cohort | Subject id. | Date | Radiography result | Specify | Other |
|-------------|-------------|------|--------------------|---------|-------|

### Listing 11.5 ECG Abnormalities

| Dose cohort | Subject id. | Date | ECG<br>Result | Specify | QT | PR | RR |
|-------------|-------------|------|---------------|---------|----|----|----|

### Listing 11.6 ECHO/MUGA results

| Dose cohort | Subject id. | Date | Result | Specify |
|-------------|-------------|------|--------|---------|

### Listing 11.7 Six-minute walk test results

| Dose cohort | Subject id. | Date | Total distance | Number of laps | Stopped or paused | Reason for stopping or pausing |
|---|---|---|---|---|---|---|

## Listing 11.8 Six-minute walk test previous medication

| Dose cohort | Subject id. | Date | Active ingredient | Admin.<br>hour | Admin.<br>minuts | Dose |
|---|---|---|---|---|---|---|

## Listing 11.9 Six-minute walk test. Supplementary oxygen during the test

| Dose cohort | Subject id. | Supplementary oxygen needed? | Flow type | Flow type specify | Flow |
|---|---|---|---|---|---|

### Table 11.11 Patients with abnormalities in the chest X-ray (all patients)

<sup>(2)</sup> Angina; Dizziness; Pain in hip, leg or calf; None

| | | Dose ( | Cohort | |
|---|---|---|---|---|
| | 1.5 mg | 1.5 mg 2.0 mg 2.5 mg Total | | |
| | N=X | N=X | N=X | N=X |
| | | n ( | %) | |
| Patients with abnormalities in the | | | | |
| chest X-ray | | | | |

Table 11.12 Patients who presented abnormalities in the heart Ultrasound/MUGA (all patients)

| | Dose Cohort | | | |
|---|---|---|---|---|
| | 1.5 mg | 2.0 mg | 2.5 mg | Total |
| | N=X | N=X | N=X | N=X |
| | | n ( | %) | |
| Patients who presented abnormalities in the heart Ultrasound/MUGA | | | | |

Table 11.13 Multivariable analysis

| Variable | Value | DF | Estimate | Standard<br>error | Wald<br>Chi-<br>Square | Pr ><br>Chi-<br>Square | Effect | Odds<br>Ratio<br>Estimate | Lower 95%<br>Confidence<br>Limit for<br>Odds Ratio | Upper 95%<br>Confidence<br>Limit for<br>Odds Ratio |
|---|---|---|---|---|---|---|---|---|---|---|

# 12 Other analysis

Table 12.1 Vital signs

| | | Dose Cohort | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Continuous endpoints | | | 1.5 | 5 | | | | | Total |
| - | N | Mean | Median | Range | Q1 | * | <br> | <br> | |
| SBP (mmHg) | | | | | | | | | |
| DBP (mmHg) | | | | | | | | | |
| Heart rate (bpm) | | | | | | | | | |
| Temperature (°C) | | | | | | | | | |
| Respiratory rate (breaths/min) | | | | | | | | | |

<sup>\*</sup> Q3 and Std.

Table 12.2 Physical and neurological examination

| | | Dose | Cohort | |
|--------------------------|--------|--------|--------|-------|
| Endpoints | 1.5 mg | 2.0 mg | 2.5 mg | Total |
| | N=X | N=X | N=X | N=X |
| | | n ( | %) | |
| Physical examination | | | | |
| Normal | | | | |
| Abnormal | | | | |
| Neurological examination | | | | |
| Normal | | | | |
| Abnormal | | | | |

## Listing 12.1 Physical examination

| Dose cohort | Subject id. | Physical examination | Date | System | Finding |
|-------------|-------------|----------------------|------|--------|---------|

## Listing 12.2 Neurological examination

| Dose cohort | Subject id. | Neurological examination | Date | Finding |
|-------------|-------------|--------------------------|------|---------|

Table 12.3 Electrocardiogram

| ECG | | Dose Cohort | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Continuous endpoints | | 1.5 | | | | | Total | | | | | | |
| Chaponits | N | Mean | Median | Range | Q1 | * | | N | Mean | Median | Range | Q1 | * |
| QT (ms) | | | | | | | | | | | | | |
| PR (ms) | | | | | | | | | | | | | |
| RR (ms) | | | | | | | | | | | | | |

<sup>\*</sup> Q3 and Std.

Table 12.4 COVID-19 (PCR)

| | | Dose | Cohort | |
|---|---|---|---|---|
| COVID-19 (PCR) | 1.5 mg<br>N=X | 2.0 mg<br>N=X | 2.5 mg<br>N=X | Total<br>N=X |
| | | n ( | %) | |
| Has a PCR test been performed? | | | | |
| Yes | | | | |
| No | | | | |
| PCR result | | | | |
| Positive | | | | |
| Negative | | | | |

Listing 12.3 COVID-19 (PCR)

| Dose cohort | Subject id. | PCR test been performed | Date | Result |
|-------------|-------------|-------------------------|------|--------|

Table 12.5 COVID-19 (history and IgG serology)

| | | Dose | Cohort | |
|---|---|---|---|---|
| COVID-19 | 1.5 mg<br>N=X | 2.0 mg<br>N=X | 2.5 mg<br>N=X | Total<br>N=X |
| | n (%) | | | |
| Has the patient been diagnosed of COVID-19 since the completion of APLICOV-PC study? | | | | |
| Yes | | | | |
| No | | | | |
| Results IgG | | | | |
| Positive | | | | |
| Negative | | | | |
| Inconclusive | | | | |
| Has the patient received any COVID-19 vaccine? | | | | |
| Yes | | | | |
| No | | | | |
| Doses received | | | | |
| 1 | | | | |
| 2 | | | | |
| 3 | | | | |

## Listing 12.4 COVID-19 history

| Dose cohort | Subject id. | Diagnosed of<br>COVID-19<br>since the<br>completion<br>APLICOV-PC<br>study | Diagnosed<br>date | End infection Date | Ongoing |
|---|---|---|---|---|---|

## Listing 12.5 COVID-19 Serology SARS-CoV-2

| Dose cohort | Subject id. | Serology<br>performed | Date | Result IgG |
|-------------|-------------|-----------------------|------|------------|

Listing 12.6 Vaccination schedule

| Dose cohort | Subject id. | Vaccination | Dose | Vaccine type | Date |
|-------------|-------------|-------------|------|--------------|------|

Table 12.6 Pharmacological treatment

| Pharmacological treatment | | 1.5 mg<br>N=X | | 2.0 mg<br>N=X | | 2.5 mg<br>N=X | | Total<br>N=X | |
|---|---|---|---|---|---|---|---|---|---|
| | | | % | N | % | N | % | N | % |
| | Has the patient received any pharmacological treatment? | | | | | | | | |
| ATC1 | ATC2 | | | | | | | | |
| | ATC2 | | | | | | | | |
| ATC1 | ATC2 | | | | | | | | |

Listing 12.7 Pharmacological treatment

| Dose cohort | Subject id. | Active ingredients | Start<br>date | End Date | Ong. | Duration | Dose | (*) |
|---|---|---|---|---|---|---|---|---|

<sup>\*</sup> Units, Frequency, Administration route and Indication.

Table 12.7 Summary of Adverse Events

| 2 | 1.5 mg<br>N=X | | 2.0 mg<br>N=X | | 2.5 mg<br>N=X | | Total<br>N=X | |
|---|---|---|---|---|---|---|---|---|
| Patients | N | %<br>% | N | %<br>% | N | %<br>% | N | % |
| Patients with AEs | | | | | | | | |
| Patients with Grade >=3 AEs | | | | | | | | |
| Patients with SAEs | | | | | | | | |

Table 12.8 Summary of AEs, regardless of relationship, by SOC and PT by dose cohort and overall

| | | Dose | Cohort | |
|---|---|---|---|---|
| MedDRA SOC | 1.5 mg | 2.0 mg | 2.5 mg | Total |
| Preferred Term | N=X | N=X | N=X | N=X |
| | n (%) | | | |
| Subjects with any AE | | | | |
| Gastrointestinal disorders | | | | |
| Abdominal pain | | | | |
| General disorders and administration | n site conditions | | | |
| Asthenia | | | | |
| Chest discomfort | | | | |

Each patient reported once per Preferred Term (PT);

Table 12.9 Summary of AEs, regardless of relationship by SOC and PT by grade and overall. Worst grade per patient. (Dose 1.5 / 2 / 2.5 mg and total)

| AFa | A.F. | | G1 ( | | G2 | | G3 | | | | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|
| AEs | | N | % | N | % | N | % | N | % | N | % |
| Gastrointestinal disorders | Abdominal pain | | | | | | | | | | |

## Listing 12.8 All adverse events

| Dose<br>cohort | Subject id. | Age | SOC | PT | Serious adverse events | Relationship | Grade | Onset date | End<br>date |
|---|---|---|---|---|---|---|---|---|---|

Table 12.10 APLICOV - Patient description

| | | Dose | Cohort | |
|------------------------------------|--------|--------|--------|-------|
| | 1.5 mg | 2.0 mg | 2.5 mg | Total |
| | N=X | N=X | N=X | N=X |
| Age, median (range) years | | | | |
| Gender, % male | | | | |
| Median (range) time from symptom | | | | |
| onset to first administration, | | | | |
| days | | | | |
| Number of comorbidities, n (%) | | | | |
| None | | | | |
| One | | | | |
| Two or more | | | | |
| Comorbidities, n (%) | | | | |
| Cardiac disease | | | | |
| Kidney disease | | | | |
| Liver disease | | | | |
| Lung disease (COPD) | | | | |
| Asthma | | | | |
| Diabetes | | | | |
| Hypertension | | | | |
| Obesity | | | | |
| Clinical status at baseline, n (%) | | | | |
| Mild COVID-19 infection | | | | |
| Moderate COVID-19 infection | | | | |
| Severe COVID-19 infection | | | | |
| Vital signs, median (range) | | | | |
| Body temperature, °C | | | | |
| Systolic blood pressure, mmHg | | | | |
| Diastolic blood pressure, mmHg | | | | |
| Heart rate, bpm | | | | |
| Respiratory rate, bpm | | | | |
| SpO <sub>2</sub> at room air, % | | | | |
| On oxygen at baseline, n (%) | | | | |

| | | Dose ( | Cohort | |
|----------------------------------------|--------|--------|--------|-------|
| | 1.5 mg | 2.0 mg | 2.5 mg | Total |
| | N=X | N=X | N=X | N=X |
| Laboratory parameters, median (range) | | | | |
| WBC, x10 <sup>9</sup> /L | | | | |
| Platelet count, x10 <sup>9</sup> /L | | | | |
| Lymphocytes, x10 <sup>9</sup> /L | | | | |
| Serum creatinine, µmol/L | | | | |
| ALT, x ULN | | | | |
| AST, x ULN | | | | |
| LDH, x ULN | | | | |
| GGT, x ULN | | | | |
| CPK, x ULN | | | | |
| Ferritin (ng/mL) | | | | |
| D-dimer (ng/mL) | | | | |
| C-reactive protein (mg/L) | | | | |
| log <sub>10</sub> viral load, | | | | |
| median (range) copies/mL | | | | |
| Days from Plitidepsin to first | | | | |
| complication | | | | |
| Days from hospital discharge to first | | | | |
| complication | | | | |
| Time from Plitidepsin first-dose to E- | | | | |
| APLICOV inclusion (month) | | | | |

## (\*) Further covariates could be added upon request

Table 12.11 APLICOV - Patient description by severity of disease

| | | Dose ( | Cohort | |
|------------------------------------|------|----------|--------|-------|
| | Mild | Moderate | Severe | Total |
| | N=X | N=X | N=X | N=X |
| Age, median (range) years | | | | |
| Gender, % male | | | | |
| Median (range) time from symptom | | | | |
| onset to first administration, | | | | |
| days | | | | |
| Number of comorbidities, n (%) | | | | |
| None | | | | |
| One | | | | |
| Two or more | | | | |
| Comorbidities, n (%) | | | | |
| Cardiac disease | | | | |
| Kidney disease | | | | |
| Liver disease | | | | |
| Lung disease (COPD) | | | | |
| Asthma | | | | |
| Diabetes | | | | |
| Hypertension | | | | |
| Obesity | | | | |
| Clinical status at baseline, n (%) | | | | |
| Mild COVID-19 infection | | | | |
| Moderate COVID-19 infection | | | | |
| Severe COVID-19 infection | | | | |
| Vital signs, median (range) | | | | |
| Body temperature, °C | | | | |
| Systolic blood pressure, mmHg | | | | |

| | Dose Cohort | | | |
|---|---|---|---|---|
| | Mild | Moderate | Severe | Total |
| | N=X | N=X | N=X | N=X |
| Diastolic blood pressure, mmHg | | | | |
| Heart rate, bpm | | | | |
| Respiratory rate, bpm | | | | |
| SpO <sub>2</sub> at room air, % | | | | |
| On oxygen at baseline, n (%) | | | | |
| Laboratory parameters, median (range) | | | | |
| WBC, x10 <sup>9</sup> /L | | | | |
| Platelet count, x10 <sup>9</sup> /L | | | | |
| Lymphocytes, x10 <sup>9</sup> /L | | | | |
| Serum creatinine, µmol/L | | | | |
| ALT, x ULN | | | | |
| AST, x ULN | | | | |
| LDH, x ULN | | | | |
| GGT, x ULN | | | | |
| CPK, x ULN | | | | |
| Ferritin (ng/mL) | | | | |
| D-dimer (ng/mL) | | | | |
| C-reactive protein (mg/L) | | | | |
| log <sub>10</sub> viral load, | | | | |
| median (range) copies/mL | | | | |
| Days from Plitidepsin to first | | | | |
| complication Days from hospital discharge to first | | | | |
| complication | | | | |
| Time from Plitidepsin first-dose to E-<br>APLICOV inclusion (month) | | | | |

Table 12.12 Laboratory parameters

| ECG | Dose Cohort | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Continuous | 1.5 | | | | | | Total | | | | | | |
| endpoints | | | | | | | | | | | | | |
| | N | Mean | Median | Range | Q1 | * | | N | Mean | Median | Range | Q1 | * |
| Hematology parameters | | | | | | | | | | | | | |
| Coagulation parameters | | | | | | | | | | | | | |
| Biochemistry parameters | | | | | | | | | | | | | |

<sup>\*</sup> Q3 and Std.

Hematology: Basophils, Eosinophils, Hematocrit, Hemoglobin, Leukocytes, Lymphocytes, Monocytes, Neutrophils, Platelets.

Biochemistry: ALT, AST, Albumin, BUN, C-Reactive Protein, CPK, Calcium, Creatinine, Ferritin, GGT,

Glomerular filtrate, Glucose, LDH, Magnesium, Phosphatase alkaline, Potassium, Sodium, Total bilirubin, Troponin I, Troponin T. Coagulation: Activated Partial Thromboplastin, D-Dimer, INR, Prothrombin Time

# 13 Other Listings

Listing 13.1 Hematological laboratory parameters

| Dose | Subject id. | Date | Parameter | Value | Units | (*) |
|------|-------------|------|-----------|-------|-------|-----|

<sup>\*</sup>Range, grade, result and clinically significant

Listing 13.2 Coagulation laboratory parameters

| Dose | Subject id. | Date | Parameter | Value | Units | (*) |
|------|-------------|------|-----------|-------|-------|-----|

<sup>\*</sup>Range, grade, result and clinically significant

Table 13.3 Biochemical laboratory parameters

| Dose | Subject id. | Date | Parameter | Value | Units | (*) |
|------|-------------|------|-----------|-------|-------|-----|

<sup>\*</sup>Range, grade, result and clinically significant

## 14 ICH Listings

Following ICH E-3 guideline, patient listings will be performed.

- 16.2.1 Discontinued Patients
- 16.2.2 Protocol Deviations
- 16.2.3 Patients Not Included in the Efficacy Analysis
- 16.2.4 Demographic Data
- 16.2.5 Compliance and/or Drug Concentration Data Not applicable as data will not be collected
- 16.2.6 Individual Efficacy Response Data Not applicable as data will not be collected
- 16.2.7 Adverse Event Listing (each patient)
   16.2.8 Listing of Individual Laboratory Measurements by Patient

## 15 History of changes

Clarifications and modifications have been added to the SAP v2.0 on date 17 Nov 2022.

All changes are included due to improved medical compression of this study.

The following tables have been added:

- Table 11.1.2 End points I by Severity of disease
- Table 11.2.1.2 Summary of post-COVID-19 complications, regardless of relationship, by severity of disease and overall. Worst per patient
- Listing 11.1.2 Post-COVID-19 complications (related to study disease)
- Table 11.10.2 Six-minute walk test (II) by severity of disease
- Table 12.10 APLICOV Patient description
- Table 12.11 APLICOV Patient description by severity of disease
- Table 12.12 Laboratory parameters

"I have read this statistical analysis plan and confirm that to the best of my knowledge it accurately describes the analytical methods".

## Reviewers:



## Approver:

